CLINICAL TRIAL: NCT04610125
Title: Clinical Trial of CAR-T in the Treatment of Relapsed and Refractory Hematopoietic and Lymphoid Tissue Tumors in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Children CAR-T
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-08

CONDITIONS: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — CF regimen; Leukapheresis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auto CAR-T (Experimental): Patients will be treated with Auto CAR-T cells
  Interventions: Biological: Auto CAR-T; Drug: Cyclophosphamide,Fludarabine; Procedure: Leukapheresis

INTERVENTIONS:
Biological: Auto CAR-T — Biological: Auto CAR-T
Drug: Cyclophosphamide,Fludarabine — Drug: Cyclophosphamide,Fludarabine
Procedure: Leukapheresis — Leukapheresis

SUMMARY:
This is an open, single-arm, prospective，clinical study to evaluate efficacy and safety of Auto CAR-T cell injection in the treatment of recurrent or refractory Hematopoietic and Lymphoid Tissue Tumors in Children

DETAILED DESCRIPTION:
A single car consists of scFv, hinge region, transmembrane region, costimulatory domain and zeta subunit of CD3.Prior to CAR-T cell infusion, the patients will be subjected to preconditioning treatment. After CAR-T cell infusion, the patients will be evaluated for adverse reactions and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent and be willing and able to comply with the visit, treatment regimen, laboratory examination and other requirements of the study as stipulated in the trial flow chart;
2. Patients with relapsed and refractory hematopoiesis and lymphoid tissue tumors confirmed by clinical diagnosis;
3. Age: 1-18 years (including boundary value), both male and female;
4. Subjects with Lansky score ≥ 50;
5. The results of treatment-related antigens were positive;
6. The expected survival time is more than 3 months from the date of signing the informed consent.

Exclusion Criteria:

1. Severe cardiac insufficiency and left ventricular ejection fraction < 50%;
2. He had a history of severe lung function damage;
3. Combined with other advanced malignant tumors;
4. Severe infection was found and could not be effectively controlled;
5. With metabolic diseases (except diabetes mellitus);
6. Combined with severe autoimmune disease or congenital immunodeficiency;
7. Untreated active hepatitis (hepatitis B, defined as positive HBsAg, HBV-DNA ≥ 500 IU / ml and abnormal liver function; hepatitis C, defined as hepatitis C antibody [HCV AB] positive, HCV-RNA higher than the detection limit of the analysis method and abnormal liver function) or combined with hepatitis B and hepatitis C co infection;
8. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), or syphilis infection;
9. Severe allergy history of biological products (including antibiotics);
10. Patients with acute graft-versus-host reaction (GVHD) after one month of discontinuation of immunosuppressants were still present;
11. The presence of other serious physical or mental illness or laboratory abnormalities that may increase the risk of participating in the study, or interfere with the results of the study, and patients considered unsuitable for the study by the investigator.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2023-06-22 (Estimated); Study Completion 2025-06-22 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Remission Rate | 3 months post CAR-T cells infusion
  Remission Rate including complete remission(CR)、partial response(PR)、No remission(NR)、progressive disease(PD)

SECONDARY OUTCOMES:
Efficacy:duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
Efficacy: progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time

CONTACTS AND LOCATIONS:
Overall Officials: Lian Jiang, MD, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Pediatric hematology, Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei, China